CLINICAL TRIAL: NCT06539351
Title: A Pilot Study to Finetune Skin Processing Procedures in Recent Vaccinees, Prior to GeKoSkimm Study Initiation
Brief Title: A Pilot Study to Finetune Skin Processing Procedures in Recent Vaccinees, Prior to GeKoSkimm Study Initiation (GeKoSkimm-pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1777/24A
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Yellow Fever
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Intervention Model Description: Pilot study to optimize sample processing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Other)
  Interventions: Other: Skin biopsy

INTERVENTIONS:
Other: Skin biopsy — 4mm skin punch biopsy

SUMMARY:
This pilot study aims to optimize the sample processing techniques for collecting and analyzing skin biopsies obtained from individuals routinely vaccinated against yellow fever. By addressing logistical challenges early, risks will be mitigated and the main study's efficiency will be enhanced.

In order to do so, 15 participants will be identified at the ITM polyclinic after receiving a yellow fever vaccination. Participants will be invited to one study visit at the ITM Clinical Trial Site (CTS) 28 days after vaccination to collect blood samples, skin punch biopsies and a minimally-invasive microbiopsy at the site of vaccination. To investigate the ideal location for the skin punch biopsies, participants will be divided in 3 groups; in the first 5 participants the biopsies will be taken directly on the vaccination site, for the next 5 participants, the biopsies will be taken at +/- 3 cm distance from the vaccination site, and for the last five participants, the biopsies will be taken at +/- 10 cm distance from the vaccination site.

ELIGIBILITY:
Inclusion Criteria:

* BMI lower than 30kg/m²
* Able and willing to provide written informed consent
* Having received a yellow fever vaccination 28 days (+2 or -2 days) ago

Exclusion Criteria:

* Any confirmed or suspected immunosuppressive or immunodeficient state (incl. cancer); asplenia; recurrent severe infections and use of immunosuppressant medication within the last 6 months prior to recruitment, except topical or short-term oral steroids
* History of bleeding disorder (e.g., factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following venipuncture
* Any other significant disease, disorder, planned surgery, or finding which may significantly affect the ability of the volunteer to participate in the study
* Tendency to keloid (scar) formation in response to skin damage

Skin diseases at the biopsy or vaccination site

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Optimize sample processing for optimal cell yield | 1 day
  To test the sample processing flow. This involves evaluating the efficiency and practicality of sample collection, preservation, and analysis protocols to ensure optimal cell yield.

SECONDARY OUTCOMES:
Absolute number of YFC-specific TRM cells per skin biopsy | 1 day
  Using different skin dissociation protocols, the absolute number of YFV-specific TRM cells that can be isolated out of 4mm punch biopsy skin samples, as determined by flow cytometry.
percentage of YFC-specific TRM cells per skin biopsy | 1day
  Using different skin dissociation protocols, the percentage of YFV-specific TRM cells that can be isolated out of 4mm punch biopsy skin samples, as determined by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Adriaensen, Prof, Principal Investigator — Coordinating Investigator
Locations (1):
- Clinical Trial Site ITM, Antwerp, Belgium